CLINICAL TRIAL: NCT03908021
Title: The Salivary Microbiome in Children With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0714-18-HMO
Record Dates: First submitted 2019-04-01; First posted 2019-04-09 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-01

CONDITIONS: Type1 Diabetes Mellitus
Keywords: diabetes mellitus; children; microbiome
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with type 1 diabetes mellitus: Saliva from 50 children ages 5 to 15 years old who had been diagnosed with type 1 diabetes mellitus and are followed at the Pediatric Endocrinology Clinic, Hadassah University Hospital Mt. Scopus and Ein Kerem, Jerusalem, Isreal,
  Interventions: Diagnostic Test: Microbiome analysis and 16S rRNA gene-based analysis
- Control: 50 healthy children, preferably their siblings, matched in age and gender.
  Interventions: Diagnostic Test: Microbiome analysis and 16S rRNA gene-based analysis

INTERVENTIONS:
Diagnostic Test: Microbiome analysis and 16S rRNA gene-based analysis — microbial DNA is extracted from the saliva and 16s library is prepared for sequencing.

SUMMARY:
Aims: To profile the oral microbiome of children with type 1 diabetes mellitus, and to compare it to healthy children while taking into account other aspects of the oral environment.

Research: exploring the differences between oral microflora of children with type 1 diabetes mellitus and control healthy children using salivary microbiome. The investigators will furthermore intend to analyze the differences of salivary flow rate, pH, glucose, calcium, inorganic phosphate and urea between the two groups.

DETAILED DESCRIPTION:
Saliva from 50 children ages 5 to 15 years old who had been diagnosed with type 1 diabetes mellitus and are followed at the Pediatric Endocrinology Clinic, Hadassah University Hospital Mt. Scopus and Ein Kerem, Jerusalem, Isreal, will be compared to 50 healthy children, preferably their siblings, matched in age and gender. Each patient or their legal guardian will sign an informed consent to participate in the study. The investigators will request a permission to access the medical records of the patients. Data will be collected from patient medical history. The investigators will measure salivary flow rate, pH and glucose, salivary Calcium, inorganic phosphate and urea and perform microbiome analysis and 16S rRNA gene-based analysis comparing children with diabetes to healthy children.

ELIGIBILITY:
Inclusion Criteria:

• Children with type 1 diabetes mellitus

Exclusion Criteria:

* Children Unable to give saliva sample
* Children On antibacterial medicaments

Ages: 5 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Saliva from 50 children ages 5 to 15 years old who had been diagnosed with type 1 diabetes mellitus and are followed at the Pediatric Endocrinology Clinic, Hadassah University Hospital Mt. Scopus and Ein Kerem, Jerusalem, Isreal, will be compared to 50 healthy children, preferably their siblings, matched in age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
profile the oral bacteria related to caries and periodontal disease of children with type 1 diabetes mellitus | 1 year
  Profile salivary microbiota in diabetic children followed by bioinformatics analyses and combining the data with the alteration in caries index, medications, state of the disease and salivary components to give a list of specific bacteria that are different in the diabetic child from healthy population.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No